CLINICAL TRIAL: NCT02759653
Title: Norwegian Carotid Plaque Study (NOR-PLAQ). Advanced Neurosonology in Acute Ischemic Stroke
Brief Title: Norwegian Carotid Plaque Study
Acronym: NOR-PLAQ
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/1217
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2016-08

CONDITIONS: Ischemic Stroke; Carotid Artery Disease; Embolic Stroke
MeSH Terms: conditions — Ischemic Stroke; Carotid Artery Diseases; Embolic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Symptomatic: Symptomatic carotid artery disease
- Asymptomatic: Asymptomatic carotid artery disease

SUMMARY:
BACKGROUND: In 30-40% the cause of ischemic stroke remains undetermined. Most likely, this category hides an additional number of strokes caused by artery-to-artery embolisms due to unidentified atherosclerotic disease, or caused by cardioembolism. Both types are associated with a high risk of recurrent ischemic events and multiple cerebral infarctions.

Large-artery atherosclerosis of the brain-supplying arteries is the assumed underlying cause in 10 to 15% of ischemic stroke, mostly deriving from the extracranial carotid artery. Carotid intima-media thickness (cIMT) measured by 2-dimensional (2D) B-mode ultrasonography and estimation of the overall atherosclerotic plaque burden aids future risk prediction. Arterial wall changes, artery caliber variations, degree of stenosis, local hemodynamic alterations and certain plaque characteristics are important for the evaluation of plaque vulnerability and vascular risk stratification. Transcranial Doppler monitoring (TCDM) is a non-invasive bedside examination eligible for detection of microemboli in the human cerebral circulation.

HYPOTHESIS: Atherosclerotic stenosis and plaque characteristics can be more accurately assessed by the combination of routine 2D ultrasound, contrast enhanced ultrasound (CEUS), and 3-dimensional (3D) ultrasound. TCDM, CEUS and 3D visualization of the carotid plaque improve the differentiation of stroke etiology and quantification of plaque vulnerability, and aid the prediction of future risk for cerebrovascular events in the individual patient.

AIMS: Assessment of prevalence and frequency of Microemboli signals (MES) in unselected patients with cerebral ischemia, the influence of antithrombotic drugs on MES, and the relationship between MES and recurrent stroke or Transient ischemic attack (TIA).

Categorization of atherosclerotic carotid artery disease by use of routine and advanced neurosonographic techniques combined with anamnestic and clinical data.

Development of a visualization solution tailored for 3D visualization of carotid arteries and semi-automatic plaque segmentation.

DETAILED DESCRIPTION:
* Standardized questionnaire
* Extracranial and transcranial duplexsonography
* Extracranial contrast-enhanced ultrasound
* Extracranial 3D-ultrasound
* Transcranial Doppler monitoring
* Clinical work-up incl. radiological and cardiological procedures, scoring etc

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic carotid artery disease
* Asymptomatic carotid artery disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic and asymptomatic carotid artery disease admitted to the Dept. of Neurology at Haukeland University Hospital, Bergen/ Norway
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Ischemic stroke or TIA documented by Medical record | 3 months

SECONDARY OUTCOMES:
Any arterial event documented by Medical record (composite) | 3 months
  Ischemic stroke, TIA, Coronary artery disease, Myocardial infarction, Peripheral arterial disease

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Aarli SJ, Thomassen L, Waje-Andreassen U, Logallo N, Kvistad CE, Naess H, Fromm A. The Course of Carotid Plaque Vulnerability Assessed by Advanced Neurosonology. Front Neurol. 2021 Aug 20;12:702657. doi: 10.3389/fneur.2021.702657. eCollection 2021. PMID 34489850